CLINICAL TRIAL: NCT04038333
Title: Influenza Vaccination Among Three Recommended Groups in China: Economic Burden, Vaccine Hesitancy, Discrete Choice Experiment, Immunization Records, Willingness to Pay and Financing Strategies
Brief Title: Financing Strategies of Influenza Vaccination in China
Status: Completed | Type: Observational
Sponsor: Peking University (Other)
Collaborators: Centers for Disease Control and Prevention, China (Other Government); Fudan University (Other); Shandong University (Other)
Responsible Party: Principal Investigator, Hai Fang, Professor, Peking University
Other Study IDs: IRB00001052-19076
Record Dates: First submitted 2019-07-22; First posted 2019-07-30 (Actual); Last update posted 2022-01-24 (Actual); Status verified 2022-01

CONDITIONS: Influenza Vaccines; Influenza, Human; Cost of Illness; Health Knowledge, Attitudes, Practice; Immunization Programs
MeSH Terms: conditions — Influenza, Human; Behavior

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Children: Interviewees are parents or grandparents of children aged between 6 to 59 months.
  Interventions: Other: No intervention
- Elderly: Interviewees are the elderly aged 60 years old or above.
  Interventions: Other: No intervention
- Chronic disease patients: Interviewees are adult patients with chronic diseases aged below 60 years old.
  Interventions: Other: No intervention
- Vaccination and health care personnel: Interviewees are vaccination and health care personnel in each study site.
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — This is an observational study without any interventions.

SUMMARY:
This trial focuses on influenza vaccination among three recommended groups in China. Data concerning the economic burden of influenza-like illness (ILI), vaccine hesitancy, discrete choice experiment, immunization records and willingness to pay for vaccines will be collected via questionnaires, and the financing strategies of influenza vaccines in China will be further analyzed. Besides, the knowledge, attitude/belief and practice (KAP) of medical staff will also be asked in a supplementary questionnaire.

DETAILED DESCRIPTION:
This trial focuses on influenza vaccination among three recommended groups in China, including children (aged between 6 to 59 months), the elderly (aged 60 years old or above), and adult patients with chronic diseases (aged below 60 years old).

The questionnaires will collect data on the economic burden of influenza-like illness (ILI), vaccine hesitancy, discrete choice experiment, immunization records and willingness to pay for vaccines, and the financing strategies of influenza vaccines in China will be further analyzed accordingly.

Besides the three recommended groups, vaccination and health care personnel will also be asked about their knowledge, attitude/belief and practice (KAP) in a supplementary questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* (For children group) children aged between 6 to 59 months.
* (For the elderly group) the elderly aged 60 years old or above.
* (For chronic disease patient group) adult patients with chronic diseases aged below 60 years old.
* (For medical staff) general practitioners and vaccination staff.
* Interviewees with informed consent.

Exclusion Criteria:

* Those cannot be surveyed for physical reasons.
* Those with communication barriers.
* Those who do not agree to participate in the survey.

Min Age: 6 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Three recommended groups for influenza vaccination in China, including children (aged between 6 to 59 months), the elderly (aged 60 years old or above), and adult patients with chronic diseases (aged below 60 years old); Vaccination and health care personnel in each study site.
Sampling Method: Probability Sample
Enrollment: 13542 (Actual)
Dates: Start 2019-08-01 (Actual); Primary Completion 2019-10-30 (Actual); Study Completion 2021-03-10 (Actual)

PRIMARY OUTCOMES:
economic burden of influenza-like illness (ILI) | 2019.08-2019.09
  Questions were designed in the questionnaire to ask the economic burden of influenza-like illness (ILI), including direct and indirect costs. Specifically, direct costs include inpatient cost (both out-of-pocket and reimbursed, range 0-100,000), hospitalization cost (both out-of-pocket and reimbursed, range 0-500,000), drug cost (both out-of-pocket and reimbursed, range 0-100,000), transportation cost (range 0-100,000), accommodation cost range (0-100,000) and food cost (range 0-100,000). Indirect cost include missed working days of the patients and their relatives/friends.
willingness to pay | 2019.08-2019.09
  Questions were designed in the questionnaire to ask interviewees' willingness to pay for influenza vaccination. A value between 0 and 150 RMB will be randomly generated, and ask the respondent whether he or she is willing to pay for influenza vaccination. For example, one is asked "Would you like pay 102 for influenza vaccination?" If the answer is "Yes", then he or she will be asked "Would you like pay 112 for influenza vaccination?" If the answer is "No", then he or she will be asked "Would you like pay 92 for influenza vaccination?" The willingness to pay is then settled and recorded. Moreover, the proportion of vaccination cost paid by individuals will be asked (if others will be paid by health insurance and the government).

SECONDARY OUTCOMES:
vaccine hesitancy and immunization records | 2019.08-2019.09
  Immunization records of children were collected. Questions were designed in the questionnaire to evaluate the degree of vaccine hesitancy of interviewees. Respondents will be asked abound their confidence, convenience and complacency about vaccination of different vaccines (include influenza, Hib, PCV, Rota and chickenpox), so as to further explore the influencing factors of people's vaccination behaviors.
financing strategies | 2019.08-2019.09
  Financing strategies will be further discussed according to literature review, government reports, and the results of willingness to pay.
  Literature review will be done to learn about the financing strategies of influenza vaccination all over the world. Government reports on basic public health financing will be an important evidence and reference. The results of willingness to pay from the questionnaire estimate the amount (0-150) and proportion (0-100%) an individual is willing to pay for influenza vaccination.
  Combining the three information sources, a supply-demand curve can be drawn to decide the optimal financing strategies of influenza vaccine, and the cross-region inequities in China will also be taken into consideration.
discrete choice experiment | 2019.08-2019.09
  An extra questionnaire was specially designed for a small portion of randomly chosen interviewees to conduce discrete choice experiment. In the discrete choice experiment, different packages of vaccine will be given for respondents to choose from. These packages have different characteristics in terms of protection duration, vaccine cost, efficacy, safety and production place. In the experiment, participants are asked to choose one package from 10 pairs of packages (package A and package B) according to their own preferences. Their preferences (protection duration, vaccine cost, efficacy, safety and production place) will be calculated and ranked according to the experiment results.

CONTACTS AND LOCATIONS:
Overall Officials: Hai Fang, PhD, Principal Investigator — Peking University
Locations (3):
- China (3):
  - Peking University Health Science Center, Beijing, Beijing Municipality
  - Shandong University, Jinan, Shandong
  - Fudan University, Shanghai, Shanghai Municipality

IPD SHARING:
Plan to Share IPD: Undecided
It is not yet known if there will be a plan to make IPD available.

REFERENCES:
- [Result] Hou Z, Jie Chang, Yue D, Fang H, Meng Q, Zhang Y. Determinants of willingness to pay for self-paid vaccines in China. Vaccine. 2014 Jul 31;32(35):4471-4477. doi: 10.1016/j.vaccine.2014.06.047. Epub 2014 Jun 23. PMID 24968160
- [Result] Rajamoorthy Y, Radam A, Taib NM, Rahim KA, Munusamy S, Wagner AL, Mudatsir M, Bazrbachi A, Harapan H. Willingness to pay for hepatitis B vaccination in Selangor, Malaysia: A cross-sectional household survey. PLoS One. 2019 Apr 9;14(4):e0215125. doi: 10.1371/journal.pone.0215125. eCollection 2019. PMID 30964934
- [Result] Molinari NA, Ortega-Sanchez IR, Messonnier ML, Thompson WW, Wortley PM, Weintraub E, Bridges CB. The annual impact of seasonal influenza in the US: measuring disease burden and costs. Vaccine. 2007 Jun 28;25(27):5086-96. doi: 10.1016/j.vaccine.2007.03.046. Epub 2007 Apr 20. PMID 17544181
- [Result] Putri WCWS, Muscatello DJ, Stockwell MS, Newall AT. Economic burden of seasonal influenza in the United States. Vaccine. 2018 Jun 22;36(27):3960-3966. doi: 10.1016/j.vaccine.2018.05.057. Epub 2018 May 22. PMID 29801998
- [Result] Salampessy BH, Veldwijk J, Jantine Schuit A, van den Brekel-Dijkstra K, Neslo RE, Ardine de Wit G, Lambooij MS. The Predictive Value of Discrete Choice Experiments in Public Health: An Exploratory Application. Patient. 2015 Dec;8(6):521-9. doi: 10.1007/s40271-015-0115-2. PMID 25618790
- [Result] Guo N, Zhang G, Zhu D, Wang J, Shi L. The effects of convenience and quality on the demand for vaccination: Results from a discrete choice experiment. Vaccine. 2017 May 15;35(21):2848-2854. doi: 10.1016/j.vaccine.2017.04.006. Epub 2017 Apr 12. PMID 28410814
- [Result] Wong CKH, Man KKC, Ip P, Kwan M, McGhee SM. Mothers' Preferences and Willingness to Pay for Human Papillomavirus Vaccination for Their Daughters: A Discrete Choice Experiment in Hong Kong. Value Health. 2018 May;21(5):622-629. doi: 10.1016/j.jval.2017.10.012. Epub 2017 Nov 15. PMID 29753361
- [Result] Larson HJ, de Figueiredo A, Xiahong Z, Schulz WS, Verger P, Johnston IG, Cook AR, Jones NS. The State of Vaccine Confidence 2016: Global Insights Through a 67-Country Survey. EBioMedicine. 2016 Oct;12:295-301. doi: 10.1016/j.ebiom.2016.08.042. Epub 2016 Sep 13. PMID 27658738
- [Result] Larson HJ, Schulz WS, Tucker JD, Smith DM. Measuring vaccine confidence: introducing a global vaccine confidence index. PLoS Curr. 2015 Feb 25;7:ecurrents.outbreaks.ce0f6177bc97332602a8e3fe7d7f7cc4. doi: 10.1371/currents.outbreaks.ce0f6177bc97332602a8e3fe7d7f7cc4. PMID 25789200
- [Result] Larson HJ, Jarrett C, Schulz WS, Chaudhuri M, Zhou Y, Dube E, Schuster M, MacDonald NE, Wilson R; SAGE Working Group on Vaccine Hesitancy. Measuring vaccine hesitancy: The development of a survey tool. Vaccine. 2015 Aug 14;33(34):4165-75. doi: 10.1016/j.vaccine.2015.04.037. Epub 2015 Apr 18. PMID 25896384
- [Result] Melia M, O'Neill S, Calderon S, Hewitt S, Orlando K, Bithell-Taylor K, Affeln D, Conti C, Wright SB. Development of a flexible, computerized database to prioritize, record, and report influenza vaccination rates for healthcare personnel. Infect Control Hosp Epidemiol. 2009 Apr;30(4):361-9. doi: 10.1086/596043. PMID 19245312